CLINICAL TRIAL: NCT00658255
Title: A Randomized, Multicenter, Open-label, Active-controlled, Single-dose, 5-period, Incomplete Block, Cross-over Study to Evaluate the Relative Bronchodilating Effects of Formoterol When Administered Via Symbicort pMDI or Oxis Turbuhaler to Adults With Stable Asthma
Brief Title: Relative Bronchodilating Effects of Formoterol When Administered Via Symbicort Pressurized Metered-dose Inhaler (pMDI) or Oxis Turbuhaler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SD-039-0729; D5896C00729
Record Dates: First submitted 2008-04-01; First posted 2008-04-14 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Stable Asthma
Keywords: stable asthma; adults; formoterol; Symbicort; Oxis Turbuhaler; bronchodilation
MeSH Terms: interventions — Budesonide, Formoterol Fumarate Drug Combination; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: budesonide/formoterol
- 2 (Active Comparator)
  Interventions: Drug: formoterol

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: formoterol
  Other Names: Oxis Turbuhaler
  Arms: 2

SUMMARY:
The purpose of this study is to compare the therapeutic effects of formoterol in Symbicort with formoterol in Oxis Turbuhaler for the treatment of adults with stable asthma.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of asthma and baseline lung function tests as determined by the protocol
* Required and received treatment with inhaled corticosteroids within timeframe and doses specified in the protocol

Exclusion Criteria:

* Severe asthma
* Has required treatment with any non-inhaled corticosteroids within previous 4 weeks, has sensitivity to drugs specified in protocol or requires treatment with beta-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2002-10; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Average FEV1 during 12 hours | Once a week for 5 weeks during treatment period

SECONDARY OUTCOMES:
Urine levels of formoterol in 2 different formulations | Once a week (12 hour urine collection) for 5 weeks during treatment period
Safety profiles of formoterol in 2 different formulations | Once a week for 5 weeks during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Ruff, MD, Study Director — Pharmaceutical Research & Consulting Inc; Catherine Bonuccelli, Study Chair — AstraZeneca